CLINICAL TRIAL: NCT02287285
Title: Long Term Change of GLP-1 Insulinotropic Effect After GBP Surgery
Brief Title: Determinants of Diabetes Remission After Gastric Bypass Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Blandine Laferrere (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Blandine Laferrere, Professor of Medicine, Columbia University, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO1360; 1R01DK098056-01A1 (NIH); 1F32DK113747-01A1 (NIH)
Record Dates: First submitted 2014-10-10; First posted 2014-11-10 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Gastric Bypass Surgery; Exendin9
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — exendin (9-39)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Exendin9 (Experimental): Longitudinal study of insulin secretion and sensitivity in patients with type 2 diabetes before and after gastric bypass surgery.
  Interventions: Drug: Exendin9

INTERVENTIONS:
Drug: Exendin9 — Dosed at 600 pmol/kg/min for 210 minutes.
  Other Names: Exendin(9-39)

SUMMARY:
Longitudinal study of beta cell function up to 2 years after GBP surgery. Evaluation of the role of endogenous glucagon-like peptide-1 (GLP-1).

DETAILED DESCRIPTION:
The increased prevalence of obesity and type 2 diabetes (T2DM) has resulted in a surge in the number of patients seeking surgical weight loss. Gastric bypass surgery (GBP) results in 30-40% body weight loss with resolution of T2DM in 40-80% of cases. The mechanisms by which T2DM improves after GBP are unclear. Glycemic control occurs long before significant weight loss, suggesting that the nature of the procedure, rather than the weight loss, is responsible for the T2DM improvement. Recent data have singled out the role of the gut hormones known as incretins in diabetes improvement after GBP. The current proposal will study 1) whether the short and long term change in the gut hormone incretins after GBP results in improved insulin secretion in response to the administration of oral and IV glucose, in patients with diabetes undergoing GBP surgery; 2) the factors responsible for diabetes remission - or lack of - after GBP. The investigators wish to apply our finding to define better surgical outcome on diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a wide range of T2DM (duration, treatment modalities and control, in or not in remission) and scheduled for GBP surgery
* Blood pressure is under at least moderate control <160/100 mmHg
* Patients can be on dyslipidemia medications but need fasting triglyceride < 600 mg/dl
* Patients without recent (last 6 months) history of cardiovascular disease (CVD)
* BMI > 35 and < 55 kg/m2 prior to GBP surgery

Exclusion Criteria:

* Active cancer
* Unstable angina
* Recent stroke
* Current therapy that may affect glucose metabolism such as glucocorticoids, HIV medications, etc
* Active infection
* Kidney failure
* Severe liver dysfunction
* Severe respiratory or cardiac failure
* History of allergic reaction to exendin 9-39
* History of pancreatitis, history of cholelithiasis, history of alcoholism
* Presence of high triglyceride levels (>600 ng/dl)
* Pregnancy (a pregnancy test will be done prior to enrollment and prior to each procedure in all premenopausal women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Beta Cell Sensitivity (BCS) | at 2 years post GBP surgery
  Oral glucose tolerance test (OGTT) will be used to calculate BCS Graded glucose infusion with arginine (GGI) will be used to calculate BCS

SECONDARY OUTCOMES:
Insulin Secretion Rate (ISR) after OGTT | 2 years post GBP surgery
  An oral glucose tolerance test (OGTT) will be used to estimate ISR in subjects before and up to 2 years after GBP
Insulin Secretion Rate (ISR) after GGI | 2 years post GBP surgery
  A graded glucose infusion with arginine (GGI) will be used to estimate ISR in subjects before and up to 2 years after GBP
Maximal Beta Cell Function | 2 years post GBP surgery
  The effect of a graded glucose infusion with arginine (GGI) on insulin secretion rate (ISR) will be measured in subjects before and up to 2 years after GBP

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — New York Obesity Nutrition Research Center, Columbia University
Locations (1):
- New York Obesity Research Center, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data generated from this study will be presented at national or international conferences and published in a timely fashion. All final peer-reviewed manuscripts that arise from this study will be submitted upon acceptance for publication to the digital archive NIH National Library of Medicine PubMed Central (PMC) database, according to the NIH Policy on Enhancing Public Access to Archived Publications Resulting from NIH Funded Research. Any data released for publication will be for research purposes only and will not include identifiable data on any of the participants.
Supporting Information: Study Protocol, ICF
Time Frame: Wherever applicable, fully de-identified data will be deposited to appropriate public repositories, following the Federal Health Insurance Privacy and Portability Act (HIPAA). This will occur no longer than 6 months after publications of the data generated by this record, or, 18 months after completion of the funding period, should no data had been published..
Access Criteria: contact the PI

REFERENCES:
- [Derived] Prasad M, Mark V, Ligon C, Dutia R, Nair N, Shah A, Laferrere B. Role of the Gut in the Temporal Changes of beta-Cell Function After Gastric Bypass in Individuals With and Without Diabetes Remission. Diabetes Care. 2022 Feb 1;45(2):469-476. doi: 10.2337/dc21-1270. PMID 34857533
- [Derived] Shah A, Holter MM, Rimawi F, Mark V, Dutia R, McGinty J, Levin B, Laferrere B. Insulin Clearance After Oral and Intravenous Glucose Following Gastric Bypass and Gastric Banding Weight Loss. Diabetes Care. 2019 Feb;42(2):311-317. doi: 10.2337/dc18-1036. Epub 2018 Dec 6. PMID 30523032